CLINICAL TRIAL: NCT02374060
Title: PeriOcular and INTravitreal Corticosteroids for Uveitic Macular Edema Trial
Acronym: POINT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006139; 1U10EY024527-01 (NIH)
Record Dates: First submitted 2015-02-18; First posted 2015-02-27 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-05

CONDITIONS: Macular Edema; Uveitis
MeSH Terms: conditions — Macular Edema; Uveitis | interventions — Triamcinolone Acetonide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Periocular triamcinolone 40mg (Active Comparator): Periocular triamcinolone acetonide (Kenalog), 40 mg Initial injection at Week 0
  Second injection permitted at Week 8 IF:
  * Eye does not meet the improvement definition (a 20% decrease in central subfield thickness of the macula) OR eye has a normal central subfield thickness but has cystoid spaces in the 1 mm central subfield OR ME is worse after initial improvement;
  * IOP of ≤21 or mm Hg and treatment with ≤3 IOP-lowering agents;
  Interventions: Drug: Periocular triamcinolone 40 mg
- Intravitreal triamcinolone 4mg (Active Comparator): (preservative-free preparation, Triescence at U.S. clinics; Triesence preferred at non-U.S. clinics but Kenalog allowed) (4 mg) Initial injection at Week 0
  Second injection permitted at Week 8 IF:
  * Eye does not meet the improvement definition (a 20% decrease in central subfield thickness of the macula) OR eye has a normal central subfield thickness but has cystoid spaces in the 1 mm central subfield OR ME is worse after initial improvement;
  * IOP of ≤21 or mm Hg and treatment with ≤3 IOP-lowering agents;
  Interventions: Drug: Intravitreal triamcinolone 4 mg
- Dexamethasoneintravitreal implant (Active Comparator): Dexamethasone intravitreal implant (Ozurdex) (0.7 mg) Initial injection at Week 0
  Second injection permitted at Week 12 IF:
  * Eye does not meet the improvement definition (a 20% decrease in central subfield thickness of the macula) OR eye has a normal central subfield thickness but has cystoid spaces in the 1 mm central subfield OR ME is worse after initial improvement;
  * IOP of ≤21 or mm Hg and treatment with ≤3 IOP-lowering agents;
  Interventions: Drug: Dexamethasone intravitreal implant

INTERVENTIONS:
Drug: Periocular triamcinolone 40 mg — Periocular triamcinolone acetonide, 40 mg injection may be given either by posterior sub-Tenon's approach or by the orbital floor approach, as both appear to have similar efficacy; the approach to the periocular injection will be recorded for analysis if needed.
  Other Names: Kenalog
  Arms: Periocular triamcinolone 40mg
Drug: Intravitreal triamcinolone 4 mg — Intravitreal triamcinolone acetonide, 4 mg injection procedures should be carried out under controlled aseptic conditions which include the use of sterile gloves and a sterile eyelid speculum (or equivalent). Adequate anesthesia and a broad-spectrum microbicide such as betadine, applied to the periocular skin, eyelid and ocular surface are required prior to an intravitreal injection.
  Other Names: Triescence (in U.S); Kenalog allowed at non-U.S. clinics
  Arms: Intravitreal triamcinolone 4mg
Drug: Dexamethasone intravitreal implant — • Standard preparation as described for intravitreal injections.
  Other Names: Ozurdex
  Arms: Dexamethasoneintravitreal implant

SUMMARY:
To evaluate the relative efficacy of three commonly utilized regional corticosteroids for the regional treatment of uveitic macular edema: periocular triamcinolone acetonide; intravitreal triamcinolone acetonide; intravitreal dexamethasone implant. The primary efficacy measure will be percent change in central subfield thickness as measured by OCT at 8 weeks. Participants will continue in the study for 24 weeks in order to evaluate relative effects of the 3 treatment strategies on the duration of treatment effects, requirement for additional injections, and adverse effects.

Note: The planned sample size for the POINT Trial was 267 subjects. On 17 July 2017, with 192 subjects enrolled, the Data and Safety Monitoring Committee (DSMC) reviewed the planned interim analysis and recommended that the goals of the trial could be accomplished by completing follow-up of enrolled subjects without the recruitment of additional subjects. Per the DSMC recommendations, recruitment was suspended and follow-up of enrolled subjects was completed according to the protocol.

DETAILED DESCRIPTION:
Macular edema is the most common structural complication and leading cause of visual loss in patients with uveitis. Regional injections of corticosteroids are the most frequently used treatments specifically for uveitic macular edema but there is a lack of high quality evidence to guide choice of drug (e.g., triamcinolone acetonide, dexamethasone) and route of administration (e.g. periocular, intravitreal). The question of how to approach regional treatment of uveitic macular edema is a key question for ophthalmologists treating these patients. The Periocular and Intravitreal Corticosteroids for Uveitic Macular Edema (POINT) Trial is a randomized trial designed to compare the relative efficacy of three regional corticosteroids commonly utilized for the initial regional treatment of uveitic macular edema, periocular triamcinolone (Kenalog® , Bristol-Myers Squibb Company, Princeton, NJ), intravitreal triamcinolone (Triesence™, Alcon Pharmaceuticals, Fort Worth, TX), and the intravitreal dexamethasone implant (Ozurdex®, Allergan, Irvine CA) will be conducted by the MUST Research Group clinical centers throughout the U.S. and one each in Australia and the UK. After signing informed consent and undergoing eligibility evaluation, eligible patients will be randomized to one of the three study treatments to be administered at the first study visit. Randomization is by participant, if both eyes meet eligibility requirements then both eyes receive assigned treatment. The design outcome is the percent change in central subfield macular thickness on OCT from baseline to the 8 week visit. After assessment of the primary outcome at 8 weeks, second injections and best medical judgment will be used if macular edema has not improved as follows:

Eye(s) meeting trial eligibility criteria receive initial injection of assigned treatment at P01 visit.

Second injection of assigned treatment permitted at 8 week visit for periocular triamcinolone and intravitreal triamcinolone and at 12 week visit for intravitreal dexamethasone if

* Eye does not meet the improvement definition (a 20% decrease in central subfield thickness of the macula) or
* Eye has a normal central subfield thickness but has cystoid spaces in the 1 mm central subfield or
* ME is worse after initial improvement

And the following repeat injection criterion are met:

• IOP of ≤21 or mm Hg and treatment with ≤3 IOP-lowering agents;

Eyes demonstrating no improvement or worsening of ME as measured by the central submacular thickness on OCT (at week 12 for periocular and intravitreal triamcinolone arms and at week 20 for intravitreal dexamethasone arm) are considered primary treatment non-responders.

ELIGIBILITY:
Inclusion Criteria:

Eye level inclusion criteria - at least one eye must meet all of the following conditions:

* Non-infectious anterior, intermediate, posterior or panuveitis; either active or inactive uveitis is acceptable;
* Macular edema (ME) defined as the presence of central subfield macular thickness greater than the normal range for the OCT machine being used, regardless of the presence of cysts, as assessed by study ophthalmologist;
* Best corrected visual acuity (BCVA) 5/200 or better;
* Baseline intraocular pressure > 5 mm Hg and ≤ 21 mm Hg (current use of 3 or fewer intraocular pressure-lowering medications and/or prior glaucoma surgery are acceptable);
* Baseline fluorescein angiogram that is gradable for leakage in the central subfield
* Pupillary dilation sufficient to allow OCT testing.

Exclusion Criteria:

Patient level exclusion criteria:

-History of infectious uveitis, or of scleritis, keratitis, or infectious endophthalmitis in either eye;

History of central serous retinopathy in either eye;

* For women of childbearing potential: pregnancy, breastfeeding, or a positive pregnancy test; unwilling to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for duration of trial;
* Use of oral acetazolamide or other systemic carbonic anhydrase inhibitor at baseline;
* Oral prednisone dose > 10 mg per day (or of an alternative corticosteroid at a dose higher than that equipotent to prednisone 10 mg per day) OR oral prednisone dose ≤ 10 mg per day that has not been stable for at least 4 weeks(note that if patient is off of oral prednisone at baseline (P01 visit), dose stability requirement for past 4 weeks does not apply);
* Systemic immunosuppressive drug therapy that has not been stable for at least 4 weeks;
* Known allergy or hypersensitivity to any component of the study drugs;

Eye level exclusion criteria - at least one eye that meets all inclusion criteria cannot have any of the following conditions:

* History of severe glaucoma as defined by optic nerve damage (cup/disc ratio of ≥ 0.9 or any notching of optic nerve to the rim);
* Media opacity causing inability to assess fundus or perform OCT;
* Presence of an epiretinal membrane noted clinically or by OCT that per the judgment of study ophthalmologist may be significant enough to limit improvement of ME (i.e., causing substantial wrinkling of the retinal surface)81;
* Torn or ruptured posterior lens capsule;
* Presence of silicone oil;
* Periocular or intravitreal corticosteroid injection in past 8 weeks;
* Injection of dexamethasone intravitreal implant in past 12 weeks;
* Placement of fluocinolone acetonide implant (Retisert) in past 3 years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Jabs, MD, MBA, Study Chair — Icahn School of Medicine, Noutn Sinai, New York, NY
Locations (26):
- United States (23):
  - Jules Stein Eye Institute, UCLA, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Anne Bates Leach Eye Hospital, University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - National Eye Institute, NIH, Bethesda, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - MAYO Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Duke Eye Center, Duke University, Durham, North Carolina
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Unniversity of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vitreoretinal Consultants, Houston, Texas
  - John A. Moran Eye Center, University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Royal Victorian Eye & Ear Hospital, East Melbourne, Australia
- McGill University, Montreal, Quebec, Canada
- Moorfields Eye Hospital, London, United Kingdom

REFERENCES:
- [Result] Thorne JE, Sugar EA, Holbrook JT, Burke AE, Altaweel MM, Vitale AT, Acharya NR, Kempen JH, Jabs DA; Multicenter Uveitis Steroid Treatment Trial Research Group. Periocular Triamcinolone vs. Intravitreal Triamcinolone vs. Intravitreal Dexamethasone Implant for the Treatment of Uveitic Macular Edema: The PeriOcular vs. INTravitreal corticosteroids for uveitic macular edema (POINT) Trial. Ophthalmology. 2019 Feb;126(2):283-295. doi: 10.1016/j.ophtha.2018.08.021. Epub 2018 Sep 27. PMID 30269924

RESULTS

PARTICIPANT FLOW:
Groups:
- Periocular Triamcinolone 40mg: Periocular triamcinolone acetonide (Kenalog), 40 mg Initial injection at Week 0
  Second injection permitted at Week 8 IF:
  * Eye does not meet the improvement definition (a 20% decrease in central subfield thickness of the macula) OR eye has a normal central subfield thickness but has cystoid spaces in the 1 mm central subfield OR ME is worse after initial improvement;
  * IOP of ≤21 or mm Hg and treatment with ≤3 IOP-lowering agents;
  Periocular triamcinolone 40 mg: Periocular triamcinolone acetonide, 40 mg injection may be given either by posterior sub-Tenon's approach or by the orbital floor approach, as both appear to have similar efficacy; the approach to the periocular injection will be recorded for analysis if needed.
- Intravitreal Triamcinolone 4mg: (preservative-free preparation, Triescence at U.S. clinics; Triesence preferred at non-U.S. clinics but Kenalog allowed) (4 mg) Initial injection at Week 0
  Second injection permitted at Week 8 IF:
  * Eye does not meet the improvement definition (a 20% decrease in central subfield thickness of the macula) OR eye has a normal central subfield thickness but has cystoid spaces in the 1 mm central subfield OR ME is worse after initial improvement;
  * IOP of ≤21 or mm Hg and treatment with ≤3 IOP-lowering agents;
  Intravitreal triamcinolone 4 mg: Intravitreal triamcinolone acetonide, 4 mg injection procedures should be carried out under controlled aseptic conditions which include the use of sterile gloves and a sterile eyelid speculum (or equivalent). Adequate anesthesia and a broad-spectrum microbicide such as betadine, applied to the periocular skin, eyelid and ocular surface are required prior to an intravitreal injection.
- Dexamethasoneintravitreal Implant: Dexamethasone intravitreal implant (Ozurdex) (0.7 mg) Initial injection at Week 0
  Second injection permitted at Week 12 IF:
  * Eye does not meet the improvement definition (a 20% decrease in central subfield thickness of the macula) OR eye has a normal central subfield thickness but has cystoid spaces in the 1 mm central subfield OR ME is worse after initial improvement;
  * IOP of ≤21 or mm Hg and treatment with ≤3 IOP-lowering agents;
  Dexamethasone intravitreal implant: • Standard preparation as described for intravitreal injections.
Period: Overall Study
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Started | 65 | 63 | 64
Completed | 63 | 62 | 61
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All eyes with uveitic macular edema at randomization according to assigned treatment ("as randomized")
Units Other Than Participants: Eyes with macular edema
Groups:
- Total: Total of all reporting groups
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant | Total
Number analyzed (Participants) | 65 | 63 | 64 | 192
Number analyzed (Eyes with macular edema) | 74 | 82 | 79 | 235
Age, Continuous [Median (Full Range); unit: years] | 55 [22 to 87] | 56 [18 to 86] | 55 [19 to 85] | 55 [18 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 40 | 119
  Male | 26 | 23 | 24 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 46 | 37 | 39 | 122
  Race: Hispanic | 1 | 3 | 5 | 9
  Race: Black | 11 | 19 | 17 | 47
  Race: Other | 7 | 4 | 3 | 14
Intraocular pressure [Median (Full Range); unit: mm Hg] | 14 [6 to 22] | 14 [7 to 21] | 13 [6 to 20] | 14 [6 to 22]
Visual acuity [Median (Full Range); unit: Standard letters] — Participants' visual acuity was measured by certified examiners with best refractive correction in place.Participants were challenged with reading letters on lines of the standard ETDRS eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until no more meaningful readings could be made and were scored by how many letters could be correctly identified. More letters read is associated with higher visual acuity.
  Standard letters | 68 [25 to 91] | 63 [13 to 88] | 64 [23 to 86] | 64 [13 to 91]
Retinal thickness at the center subfield [Median (Full Range); unit: um] | 438 [278 to 922] | 485 [236 to 824] | 449 [243 to 1300] | 462 [236 to 1300]
Concomitant systemic medication [Count of Participants; unit: Participants] | 24 | 23 | 23 | 70

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Baseline Central Subfield Thickness Observed at 8 Weeks
Description: The primary outcome is the change in central subfield thickness from baseline to 8 weeks measured on a relative scale as the the proportion of the baseline central subfield thickness. Values less than 1 indicate a decrease in retinal thickness with lower values indicating greater decreases. Smaller values are better.
  The time point of 8 weeks was chosen for assessment of the primary outcome because it encompasses the window for maximum benefit for all three treatment strategies. Retinal thickness was evaluated using masked assessments of OCT images.
Time Frame: At baseline and 8 weeks
Population: All eyes with uveitic macular edema at randomization according to assigned treatment ("as randomized")
Measure: Mean (99.87% Confidence Interval); unit: proportion of baseline retinal thickness
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
proportion of baseline retinal thickness | .77 [.67 to .89] | .61 [.53 to .70] | .54 [.46 to .63]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p < 0.0001, mixed effects model — Two sided type I error threshold was 0.00132 since recruitment was halted after the single pre-planned interim analysis; Ratio of the proportion of BL = 0.79, 99.87% CI 2-sided [.65 to .96] — Ratio of intravitreal over periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p < 0.0001, mixed effects model — the 2 sided type 1 error threshold was 0.000132 since recruitment was halted after the single preplanned interim analysis; Ratio of the proportion of BL = 0.69, 99.87% CI 2-sided [0.56 to 0.86] — ratio of dexamethasone over periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Non-Inferiority — The non inferiority margin was 1.16; Ratio of the proportion of BL = 0.88, 99.87% CI 2-sided [.71 to 1.08] — A mixed effects model was used to create the confidence interval for testing non-inferiority. The direction is the ratio of dexamethasone over intravitreal

2. Secondary Outcome: Proportion of Baseline Central Subfield Thickness Observed at 24 Weeks
Description: The primary outcome is the change in central subfield thickness from baseline to 24 weeks measured on a relative scale as the the proportion of the baseline central subfield thickness. Values less than 1 indicate a decrease in retinal thickness with lower values indicating greater decreases. Smaller values are better.The time point of 24 weeks was chosen to evaluate the duration of response and the need for additional injections.Retinal thickness was evaluated using masked assessments of OCT images.
Time Frame: At baseline and the 24 week visit
Population: All eyes with uveitic macular edema at randomization according to assigned treatment ("as randomized")
Measure: Mean (99.87% Confidence Interval); unit: proportion of baseline retinal thickness
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
proportion of baseline retinal thickness | 0.68 [0.59 to 0.79] | 0.64 [0.56 to 0.74] | 0.61 [0.52 to 0.71]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.35, mixed effects model — Two sided type I error threshold was 0.00132 since recruitment was halted after the single Two sided type I error threshold was 0.00132 since recruitment was halted after the single preplanned interim analysis; Ratio of the proportion of BL = 0.95, 99.87% CI 2-sided [0.77 to 1.16] — Ratio of intravitreal over periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.07, mixed effects model — [p-value comment as in outcome 1, analysis 2]; Ratio of the proportion of BL = 0.89, 99.87% CI 2-sided [0.72 to 1.10] — ratio of dexamethasone over periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Non-Inferiority — The non inferiority margin was 1.16; Ratio of the proportion of BL = 0.94, 99.87% CI 2-sided [0.77 to 1.16] — [estimate comment as in outcome 1, analysis 3]

3. Secondary Outcome: Proportion of Eyes With >= 20% Reduction in Macular Thickness (or Normalization Even if <20% Reduction) at 8 Weeks
Description: Proportion of eyes with >=20% reduction in macular thickness (or normalization of macular thickness even if there is <20% reduction) at 8 weeks.
Time Frame: Over 8 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: Proportion of eyes
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Proportion of eyes | 0.41 [0.29 to 0.52] | 0.79 [0.70 to 0.88] | 0.84 [0.74 to 0.94]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p < 0.0001, mixed effects model; Difference in proportion = 0.39, 95% CI 2-sided [0.24 to 0.53] — Intravitreal - periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p < 0.0001, mixed effects model; Difference in proportion = 0.44, 95% CI 2-sided [0.29 to 0.59] — Dexamethasone - periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.45, mixed effects model; Difference in proportion = 0.05, 95% CI 2-sided [-0.09 to 0.19] — Dexamethasone - intravitreal

4. Secondary Outcome: Proportion of Eyes With >= 20% Reduction in Macular Thickness (or Normalization Even if <20% Reduction) at 24 Weeks
Description: Proportion of eyes with >=20% reduction in macular thickness (or normalization of macular thickness even if there is <20% reduction) at 24 weeks
Time Frame: Over 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: Proportion of eyes
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Proportion of eyes | 0.61 [0.50 to 0.72] | 0.73 [0.63 to 0.83] | 0.74 [0.61 to 0.85]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.10, mixed effects model; Difference in proportion = 0.12, 95% CI 2-sided [-0.03 to 0.27] — Intravitreal - Periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.11, mixed effects model; Difference in proportion = 0.12, 95% CI 2-sided [-0.03 to 0.28] — Dexamethasone - Periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.98, mixed effects model; Difference in proportion = 0.002, 95% CI 2-sided [-0.16 to 0.16] — Dexamethasone - Intravitreal

5. Secondary Outcome: Proportion of Eyes With Resolution of Macular Edema at 8 Weeks
Description: Proportion of eyes with resolution of macular edema defined as normalization of the macular thickness (i.e., < 260 um on the standardized scale) at 8 weeks. The greater the proportion the more eyes achieved resolution of macular edema.
Time Frame: Over 8 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: Proportion of eyes
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Proportion of eyes | 0.20 [0.12 to 0.30] | 0.47 [0.34 to 0.60] | 0.61 [0.48 to 0.73]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.0005, mixed effects model; Difference in proportion = 0.27, 95% CI 2-sided [0.11 to 0.43] — Intravitreal - periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p < 0.0001, mixed effects model; Difference in proportion = 0.40, 95% CI 2-sided [0.25 to 0.56] — Dexamethasone - periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.12, mixed effects model; Difference in proportion = 0.13, 95% CI 2-sided [-0.04 to 0.30] — Dexamethasone - intravitreal

6. Secondary Outcome: Proportion of Eyes With Resolution of Macular Edema at 24 Weeks
Description: Proportion of eyes with resolution of macular edema defined as normalization of the macular thickness (i.e., <260 um on the standard scale) at 24 weeks.
Time Frame: Over 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: Proportion of eyes
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Proportion of eyes | 0.35 [0.24 to 0.47] | 0.36 [0.24 to 0.48] | 0.41 [0.28 to 0.54]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.96, mixed effects model; Difference in proportion = 0.004, 95% CI 2-sided [-0.16 to 0.17] — Intravitreal - periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.51, mixed effects model; Difference in proportion = 0.06, 95% CI 2-sided [-0.11 to 0.23] — Dexamethasone - periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.54, mixed effects model; Difference in proportion = 0.05, 95% CI 2-sided [-0.12 to 0.22] — Dexamethasone - intravitreal

7. Secondary Outcome: Change in Best-corrected Visual Acuity at 8 Weeks
Description: Mean change in best-corrected visual acuity from baseline to 8 weeks. Participants' visual acuity was measured by certified examiners with best refractive correction in place.Participants were challenged with reading letters on lines of the standard ETDRS eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until no more meaningful readings could be made and were scored by how many letters could be correctly identified. More letters read is associated with higher visual acuity.
Time Frame: Over 8 weeks of follow-up
Measure: Mean (95% Confidence Interval); unit: Standard letters
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Standard letters | 4.37 [1.86 to 6.89] | 9.70 [7.26 to 12.13] | 9.53 [7.01 to 12.05]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.003, mixed effects model; Difference in mean change from BL = 5.32, 95% CI 2-sided [1.82 to 8.82] — Intravitreal - periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.004, mixed effects model; Difference in mean change from BL = 5.16, 95% CI 2-sided [1.60 to 8.72] — Dexamethasone - periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.93, mixed effects model; Difference in mean change from BL = -0.16, 95% CI 2-sided [-3.67 to 3.34] — Dexamethasone - intravitreal

8. Secondary Outcome: Change in Best-corrected Visual Acuity at 24 Weeks
Description: Mean change in best-corrected visual acuity from baseline to 24 weeks. Participants' visual acuity was measured by certified examiners with best refractive correction in place.Participants were challenged with reading letters on lines of the standard ETDRS eye chart (5 letters per line). Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until no more meaningful readings could be made and were scored by how many letters could be correctly identified. More letters read is associated with higher visual acuity.
Time Frame: Over 24 weeks of follow-up
Measure: Mean (95% Confidence Interval); unit: Standard letters
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Standard letters | 4.07 [0.64 to 7.51] | 9.60 [6.87 to 12.34] | 9.21 [6.62 to 11.80]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.013, mixed effects model; Difference in mean change from BL = 5.53, 95% CI 2-sided [1.14 to 9.92] — Intravitreal - periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.019, mixed effects model; Difference in mean change from BL = 5.14, 95% CI 2-sided [0.84 to 9.44] — Dexamethasone - periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.84, mixed effects model; Difference in mean change from BL = -0.40, 95% CI 2-sided [-4.16 to 3.37] — Dexamethasone-intravitreal

9. Secondary Outcome: Number of Eyes With Vitreous Hemorrhage
Description: Count of eyes with vitreous hemorrhage as an immediate complication of injection.
Time Frame: During 24 weeks of follow-up
Measure: Number; unit: Eyes with uveitic macular edema
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Eyes with uveitic macular edema | 1 | 0 | 1

10. Secondary Outcome: Number of Eyes With Retinal Tear or Detachment
Description: Count of eyes with retinal tears or detachments during the course of follow-up.
Time Frame: During 24 weeks of follow-up
Measure: Number; unit: Eyes with uveitic macular edema
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Eyes with uveitic macular edema | 1 | 0 | 0

11. Secondary Outcome: Number of Eyes With Endophthalmitis
Description: Count of eyes with an occurrence of endophthalmitis
Time Frame: During 24 weeks of folllow-ip
Measure: Number; unit: Eyes with uveitic macular edema
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 82 | 79
Eyes with uveitic macular edema | 1 | 0 | 0

12. Secondary Outcome: Cumulative Proportion of Eyes With Severe Vision Loss
Description: Cumulative proportion of eyes with uveitic macular edema who experience severe vision loss (>= 15 standard letters) during the 24 weeks of follow-up.
Time Frame: During 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of eyes at 24 wks
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 81 | 78
Cumulative proportion of eyes at 24 wks | 0.11 [0.04 to 0.18] | 0.10 [0.0 to 0.22] | 0.05 [0.0 to 0.10]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.10, Regression, Cox; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.09 to 1.24] — Intravitreal/Periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.20, Regression, Cox; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.14 to 1.50] — Dexamethasone/Periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.62, Regression, Cox; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.34 to 6.26] — Dexamethasone/Intravitreal

13. Secondary Outcome: Cumulative Proportion of Eyes With an IOP Elevation of >=10 mm Hg Over Baseline
Description: Cumulative proportion of eyes with uveitic macular edema that experience an IOP elevation of >=10 mm Hg higher than the baseline level during 24 weeks of follow-up.
Time Frame: During 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of eyes at 24 wks
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 81 | 78
Cumulative proportion of eyes at 24 wks | 0.14 [0.05 to 0.22] | 0.26 [0.13 to 0.38] | 0.39 [0.20 to 0.53]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.11, Regression, Cox; Hazard Ratio (HR) = 1.92, 95% CI 2-sided [0.86 to 4.29] — Intravitreal/Periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.009, Regression, Cox; Hazard Ratio (HR) = 2.85, 95% CI 2-sided [1.30 to 6.28] — Dexamethasone/Intravitreal
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.30, Regression, Cox; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.72 to 2.81] — Dexamethasone/intravitreal

14. Secondary Outcome: Cumulative Proportion of Eyes With an IOP Elevation >=24 mm Hg
Description: Cumulative proportion of eyes with uveitic macular edema that experience elevated IOP to >=24 mm Hg during 24 weeks of follow-up.
Time Frame: During 24 weeks of follow-up
Population: As randomized
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of eyes at 24 wks
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 81 | 78
Cumulative proportion of eyes at 24 wks | 0.20 [0.09 to 0.29] | 0.30 [0.17 to 0.40] | 0.41 [0.26 to 0.53]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.09, Regression, Cox; Hazard Ratio (HR) = 1.83, 95% CI 2-sided [0.91 to 3.65] — Intravitreal/periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.007, Regression, Cox; Hazard Ratio (HR) = 2.52, 95% CI 2-sided [1.29 to 4.91] — Dexamethasone/periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.37, Regression, Cox; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.72 to 2.43] — Dexamethasone/intravitreal

15. Secondary Outcome: Cumulative Proportion of Eyes With an IOP Elevation >=30 mm Hg
Description: Cumulative proportion of eyes with uveitic macular edema that experience elevated IOP to >=30 mm Hg during 24 weeks of follow-up.
Time Frame: During 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: Cumulative proportion of eyes at 24 wks
Units Other Than Participants: Eyes with uveitis macular edema
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
Number analyzed (Participants) | 65 | 63 | 64
Number analyzed (Eyes with uveitis macular edema) | 74 | 81 | 78
Cumulative proportion of eyes at 24 wks | 0.06 [0.00 to 0.12] | 0.06 [0.01 to 0.12] | 0.04 [0.00 to 0.08]
Statistical Analysis 1: Comparison: Periocular Triamcinolone 40mg vs Intravitreal Triamcinolone 4mg; Test type: Superiority; p = 0.92, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.28 to 4.01] — Intravitreal/Periocular
Statistical Analysis 2: Comparison: Periocular Triamcinolone 40mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.65, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.16 to 3.11] — Dexamethasone/Periocular
Statistical Analysis 3: Comparison: Intravitreal Triamcinolone 4mg vs Dexamethasoneintravitreal Implant; Test type: Superiority; p = 0.53, Regression, Cox; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.16 to 2.59] — Dexamthasone/Intravitreal

ADVERSE EVENTS:
Time Frame: 24 weeks of follow-up
Arm/Group | Periocular Triamcinolone 40mg | Intravitreal Triamcinolone 4mg | Dexamethasoneintravitreal Implant
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 6/65 | 5/63 | 6/64
Other Adverse Events (participants affected / at risk) | 0/65 | 0/63 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Periocular Triamcinolone 40mg (N=65) | Intravitreal Triamcinolone 4mg (N=63) | Dexamethasoneintravitreal Implant (N=64)
Choroidal (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
injection site injury (General disorders) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
mediastinoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
bursitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Investigation (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT02374060/Prot_SAP_000.pdf